CLINICAL TRIAL: NCT02083003
Title: Polyamine-low Diet to Prevent Postoperative Pain After Cholecystectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: End of commercialization of low polyamin diet
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011/68; 2011-A01675-36 (Other: ANSM)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Surgery
Keywords: Pain; Polyamine; Cholecystectomy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyamine low-diet (Experimental): Polyamines depleted diet during the week before surgery : 2 cans per day of Polydol (oral alimentation without polyamines), associated to predefined menus low in polyamines
  Interventions: Dietary Supplement: Polyamine low-diet
- Liberal alimentation (Active Comparator): No specific alimentary diet
  Interventions: Dietary Supplement: Liberal alimentation

INTERVENTIONS:
Dietary Supplement: Polyamine low-diet
  Other Names: Poyldol plus (Nutrialys)
  Arms: Polyamine low-diet
Dietary Supplement: Liberal alimentation
  Other Names: No specific alimentary recommendation
  Arms: Liberal alimentation

SUMMARY:
It has been shown that N-methyl-D-aspartate (NMDA) receptor antagonists (such as ketamine) potentiate analgesic drug's efficacy. Polyamines are allosteric modulators of NMDA receptors. In animal studies, polyamine-free diet has shown antinociceptive properties. This research aims at evaluating analgesic properties of polyamine-low diet after laparoscopic cholecystectomy performed in an ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic cholecystectomy
* ambulatory surgery
* agreeing to follow a polyamine-low diet with Polydol plus

Exclusion Criteria:

* Pregnancy
* Contra-indication to a non-steroidal anti-inflammatory, to tramadol
* Intolerance to cow proteins
* Diabetic patients
* Poor understanding of the French language.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity for the 7 days | 7 days
  Pain intensity is evaluated by the number of tablets of Tramadol taken by the patients

SECONDARY OUTCOMES:
Pain scores measured on the day of surgery, | 12 hours
  Pain score (numerical scale from 0 to 10) measured in mid-afternoon, resting lying down, coughing and mobilization (from lying to sitting position)
frequency of impeded hospital discharge the day of surgery | 24 hours
  Failure of outpatient care (i.e. the patient cannot leave the hospital the day of surgery)
Each day pain | 7 days
  Pain scores (numerical scale from 0 to 10) assessed daily from J1 ( after surgery) to J7 in mid afternoon , lying at rest position , coughing and mobilization (from lying to sitting position) .
Quality of life | 7 days
  QLQC30 Questionnaire (version 3)
Residual pain | 30 days
  Pain score (numerical scale from 0 to 10)
Blood levels of polyamine | 2 years
  Blood samples are performed the day of surgery and at J7. The dosages will be performed when all patients will be recruited

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hopital Foch
Locations (1):
- Hôpital de la Croix Saint-Simon, Paris, Hauts de Seine, France